CLINICAL TRIAL: NCT01494441
Title: A Pilot Study of Recombinant Human Bone Morphogenetic Protein-2 and Biphasic Calcium Phosphate With or Without the TSRH® Spinal System for Posterolateral Lumbar Fusion in Patients With Symptomatic Degenerative Disc Disease
Brief Title: Pilot Study of rhBMP/BCP With or Without the TSRH® Spinal System for Posterolateral Lumbar Fusion in Patients With Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-9805
Record Dates: First submitted 2011-12-12; First posted 2011-12-19 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
Keywords: lumbar degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — recombinant human bone morphogenetic protein-2; hydroxyapatite-beta tricalcium phosphate; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- rhBMP-2/BCP (Experimental)
  Interventions: Procedure: rhBMP-2/BCP
- rhBMP-2/BCP/TSRH® Spinal System (Experimental)
  Interventions: Device: rhBMP-2/BCP/TSRH® Spinal System
- Autograft/TSRH® Spinal System (Active Comparator)
  Interventions: Device: Autograft/TSRH® Spinal System

INTERVENTIONS:
Procedure: rhBMP-2/BCP — The rhBMP-2/BCP device component consists of recombinant human Bone Morphogenetic Protein-2 ( rhBMP-2) and the biphasic calcium phosphate (BCP) carrier.
  Other Names: recombinant human Bone Morphogenetic Protein-2; biphasic calcium phosphate
  Arms: rhBMP-2/BCP
Device: rhBMP-2/BCP/TSRH® Spinal System — rhBMP-2/BCP device will be used in conjunction with the posterior spinal fixation system, the TSRH® Spinal System.
  Other Names: recombinant human Bone Morphogenetic Protein-2; biphasic calcium phosphate
  Arms: rhBMP-2/BCP/TSRH® Spinal System
Device: Autograft/TSRH® Spinal System — The control device will be autogenous bone from the iliac crest of the patient used in conjunction with the TSRH® spinal System.
  Other Names: Autograft
  Arms: Autograft/TSRH® Spinal System

SUMMARY:
The purpose of this pilot clinical trial is to evaluate both device designs (rhBMP-2/BCP and rhBMP-2/BCP/TSRH® spinal System) as methods of facilitating spinal fusion as compared to instrumented fusion with autograft in patients with symptomatic degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc diseases noted by back pain of discogenic origin,with or without leg pain, with degeneration of the disc confirmed by patient history ( e.g., pain [leg, back, or symptoms in the sciatic nerve distribution] function deficit and/or neurological deficit) and radiographic studies ( e.g., CT, MRl, X-Ray,etc.) to include one or more of the following:

   * instability (defined as angular motion > 5° and/or translation > 4 mm, based on Flex/Ext radiographs);
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration or herniation; and/or
   * facet joint degeneration.
2. Has preoperative Oswestry score > 30.
3. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding HW,1932.).
4. Requires fusion of a single level disc space from L1 to S1.
5. Is at least 18 years of age, inclusive, at the time of surgery.
6. Has not responded to non-operative treatment ( e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of at least 6 months.
7. If female of child-bearing potential, who is not pregnant or nursing, and who agrees to use adequate contraception for 16 weeks following surgery.
8. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Has primary diagnosis of a spinal disorder other than degenerative disc disease with Grade1 or less spondylolisthesis at the involved level.
2. Had previous spinal fusion surgical procedure at the involved level.
3. Require spinal fusion at more than one lumbar level.
4. Has a condition which requires postoperative medications that interfere with fusion, such as steroids.
5. Has been previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated.
6. Has presence of active malignancy.
7. Has overt or active bacterial infection, either local or systemic.
8. Is grossly obese, i.e., weight > 40% over ideal for their age and height.
9. Has fever ( temperature >101°F oral) at the time of surgery.
10. Has a documented titanium alloy allergy or intolerance.
11. Is mentally incompetent. If questionable, obtain psychiatric consult.
12. Has a Waddell Signs of Inorganic Behavior score of 3 or greater.
13. Is a prisoner.
14. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug usage.
15. Is a tobacco user at the time of surgery.
16. Has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., NSAIDS, steroids or methotrexate).
17. Has a history of autoimmune disease (Systemic Lupus Erythematosus or Dermatomyositis).
18. Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins).
19. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/BCP implantation.
20. Has received any previous exposure to any/all BMPs of either human or animal extraction.
21. Has a history of severe allergy (anaphylaxis).
22. Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers- Danlos syndrome, or osteogenesis imperfecta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1999-05; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Fusion | 24 month
  Fusion is defined as:
  1. Evidence of bridging trabecular bone.
  2. No evidence of motion as defined by: a. No more than 3mm difference in translation on the lateral flexion/extension radiographs determined by superimposing the two views, one upon the other; b. Less than 5° difference in angular motion between flexion and extension as seen on the lateral flexion/extension radiographs;
  3. Absence of radiolucent lines completely through the fusion mass.
Pain/Disability Status | 24 month
  The self-administered Oswestry Low Back pain Disability Questionnaire will be used. Success for each individual patient will be defined as pain/disability improvement postoperatively according to the following definition: Preoperative Score - Postoperative Score >= 15

SECONDARY OUTCOMES:
Neurological Status Success | 24 month
  Neurological status will be assessed preoperatively and postoperatively using a comprehensive neurological status scale. Neurological status is based on four types of measurements (sections): motor, sensory, reflexes and straight leg raise.
Hip (Donor Site) Pain | 24 month
General Health Status (SF-36) | 24 month
Pain Status (back pain, leg pain) | 24 month
Patient Satisfaction | 24 month
Patient Global Perceived Effect | 24 month
Overall Success | 24 month